CLINICAL TRIAL: NCT01163903
Title: A Phase I Study Evaluating the Proton Pump Inhibitor Pantoprazole in Combination With Doxorubicin for Advanced Cancer Patients With an Extension Cohort of Patients With Solid Tumours
Brief Title: Pantoprazole With Doxorubicin for Advanced Cancer Patients With Extension Cohort of Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DDP-IT-01
Record Dates: First submitted 2010-07-13; First posted 2010-07-16 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Advanced Solid Tumours
Keywords: Advanced solid tumours; Pantoprazole; Doxorubicin; PANTO IV; Adriamycin; no standard treatment options; dose-escalation schedule; Phase I; single-centre; open label; dose finding; recommended phase II dose; proton pump inhibitor; advanced cancer; anthracycline; gastric acid secretion
MeSH Terms: interventions — Pantoprazole; Injections; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pantoprazole and doxorubicin (Experimental)
  Interventions: Drug: pantoprazole sodium for injection; Drug: doxorubicin hydrochloride injection

INTERVENTIONS:
Drug: pantoprazole sodium for injection — Single 3-weekly doses of pantoprazole using the following dose escalation scheme for successive groups of patients: 80, 160, 240 and 320mg i.v. of pantoprazole to be given every 3 weeks, 30-60 (±5) minutes prior to doxorubicin. Treatment will be repeated on Day 1 of a 21-day cycle until radiographic or symptomatic progression or unacceptable toxicity or a maximum of 4 cycles (for patients who have received prior anthracyclines), and up to 8 cycles (for those with no prior exposure to anthracyclines).
  Other Names: Pantoprazole; PANTO IV
Drug: doxorubicin hydrochloride injection — 60 mg/m2, IV, scheduled on day 1 of every 3-week interval, 30-60 (±5) minutes after pantoprazole administration.
  Other Names: ADRIAMYCIN PFS; ADRIAMYCIN; doxorubicin hydrochloride

SUMMARY:
This is a single-centre, open label, dose finding, phase I study to determine the recommended phase II dose (RP2D) for the combination of doxorubicin and pantoprazole in patients with advanced tumours and no standard treatment options. A minimum of 3 patients will be enrolled per dose level and intra-patient dose escalation is not permitted. Once the RP2D has been identified, six additional patients with metastatic solid tumours will be treated at the RP2D to confirm its tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically proven advanced solid tumours for whom no standard anticancer therapy exists
2. Measureable and non-measureable disease are both eligible, but disease must be evaluable as defined by RECIST 1.1.
3. Patients >18 years old
4. At least 21 days since last chemotherapy regimen and/or radiotherapy
5. Recovery from all reversible adverse events of previous anticancer therapies to baseline or to grade < or =1, except for alopecia.
6. Patients must have documented evidence of disease progression on prior systemic therapy.
7. ECOG Performance Status of 0 or 1
8. Adequate cardiovascular function and no history of serious cardiac diseases (see Exclusion criteria for definition) Left ventricular ejection fraction > 50% by multi-gated nuclear angiogram
9. Patient consent must be obtained according to Institutional REB requirements. The patient must sign the consent form prior to registration.
10. Patients must be accessible for treatment and follow-up.
11. Previous Therapy

    1. Chemotherapy: Patients can have had limited exposure to prior anthracyclines defined as no more than a total dose of 240 mg/m2 of doxorubicin or 300 mg/m2 of epirubicin (e.g. as received in the AC x 4 or FEC x 3 adjuvant regimens). Patients with prior exposure to other cardiotoxic anticancer drugs (e.g. mitoxantrone) are not eligible.
    2. Radiation: Patients may have had prior radiation therapy (including that to the breast or chest wall) provided that has not exceeded 25% of the bone marrow reserve.
    3. Previous Surgery: Previous surgery is permitted provided that wound healing has occurred.
    4. Hormonal Therapy: Patients may have had prior hormonal therapy. All hormonal agents must be discontinued at least 3 weeks prior to study entry.
12. Laboratory Requirements (must be done within 7 days prior to registration)

    1. Neutrophil count (ANC) > or = 1.5 x 10^9/L
    2. Hemoglobin > or = 90 g/L
    3. Platelet count > or = 100 x 10^9/L
    4. Bilirubin <1.5 x UNL
    5. AST or ALT < or = 2 x UNL
    6. Creatinine < or = 1.5 x UNL or creatinine clearance > or = 50mL/min

Exclusion Criteria:

1. Patients who have previously received more than 240 mg/m2 doxorubicin or 300 mg/m2 epirubicin.
2. Patients receiving concurrent treatment with experimental drugs or anti-cancer therapy.
3. Patients who are receiving drugs that are known to interact with pantoprazole, including:

   1. The anti-fungal agents fluconazole, itraconazole, ketoconazole, posaconazole, voriconazole;
   2. The antiviral agents: atazanavir, delavirdine, indinavir, nelfinavir, raltegravir, saquinavir, tipranavir;
   3. The anticoagulant agents: clopidogrel, dabigatran;
   4. The immunosuppressive agent: mycophenolate
   5. The anti-inflammatory agent: mesalamine
4. Patients who are receiving oral pantoprazole or other PPI inhibitors may participate if these agents are discontinued at least 7 days before trial entry.
5. Patients with untreated brain or meningeal metastases. (MR or CT scans are not required to rule this out unless there is a clinical suspicion of CNS disease). Patients with treated and stable brain metastases are eligible providing that they have radiological evidence of disease stabilization of at least 3 months duration and are asymptomatic.
6. Patients who have a history of clinically significant cardiac disease, including:

   1. Unstable angina/ acute coronary syndrome
   2. Congestive heart failure
   3. Myocardial infarction within the past year
   4. Clinically significant arrhythmia
   5. Pericarditis or myocarditis
   6. Symptomatic valvular disease Patients with well-controlled hypertension, uncomplicated mitral valve prolapsed or other stable cardiac conditions are eligible.
7. Patients with active or uncontrolled infections or with serious illnesses or medical conditions that would not permit the patient to be managed according to the protocol.
8. Patients with a known bleeding disorder. Patients who are on stable anticoagulation with warfarin or s.c. heparin products are eligible. Patients receiving clopidogrel are excluded.
9. Patients unable or unwilling to give written, informed consent prior to study participation.
10. Women who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Determination of recommended phase II dose (RP2D) of pantoprazole given with doxorubicin at 60mg/m2 | Treatment until documented progression or up to 8 21-day cycles (4 cycles if prior anthracyclines received). All patients followed for late toxicities, every 3 months for 1 year or until all drug related toxicities are resolved/become unrelated.
  To determine the recommended phase II dose (RP2D) of pantoprazole given with doxorubicin at 60mg/m2 when administered to adult patients with advanced solid tumours.

SECONDARY OUTCOMES:
Characterize the safety and tolerability of the combination by determining dose-limiting toxicities (DLTs). Toxicities evaluated and graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. | Treatment until documented progression or up to 8 21-day cycles (4 cycles if prior anthracyclines received). All patients followed for late toxicities, every 3 months for 1 year or until all drug related toxicities are resolved/become unrelated.
  Three or 6 patients will be treated per cohort for at least one cycle (21 days per cycle). If two patients experience DLTs, then accrual will stop at that level, and the next lower dose level in which six patients have been treated with no or only 1 DLT will be declared the RP2D. Once the RP2D has been identified, six additional patients will be treated at the RP2D to confirm its safety and tolerability. Patients will be assessed for toxicities using the overall safety profile as per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Assess the preliminary anti-tumour activity of the doxorubicin/pantoprazole by combination in patients with advanced solid tumours, by evaluating tumour response rate. | Radiologic evaluation (CT scan of chest, abdomen and pelvis) performed every 9 weeks
  Response Evaluation Criteria in Solid Tumours (RECIST) will be used to determine radiological tumour response for measurable disease and disease progression. Changes in only the largest diameter (unidimensional measurement) of the tumour lesions are used in the RECIST criteria. Any radiological change should be confirmed using a second follow-up scan, 6 or more weeks later. For response there must be no new lesions and no evidence of progression of non-measurable lesions.
Evaluate the pharmacokinetics of doxorubicin and pantoprazole when given in combination by collecting venous blood samples at various timepoints throughout study drug administration. | Blood samples just before and at the end of pantoprazole and doxorubicin administration, and at 1, 2, 4, 8, 24, 48 and 72 hours after (first or second) drug administration for evaluation of serum levels of doxorubicin and pantoprazole
Evaluate (in selected patients with lesions amenable to biopsy) the influence of pantoprazole on distribution of doxorubicin in tumour tissue. Tumour tissue extracted after administration of doxorubicin/pantoprazole. | Tumour biopsy within 24-48h after administration of doxorubicin (in consenting patients with disease amenable to biopsy)
  Two cores of tumour tissue will be extracted within 24-48 hours of administration of doxorubicin and pantoprazole;1 core will be fixed for routine pathological examination and the 2nd will be fresh frozen. The latter will be sectioned in the experimental pathology laboratory and will be stained with antibodies which recognize tumour blood vessels and regions of hypoxia. Distribution of doxorubicin (which is fluorescent) in relation to the blood vessels in tumours, and in relation to hypoxic regions, will then be quantified using immunohistochemistry at an advanced optical microscopy facility.

CONTACTS AND LOCATIONS:
Overall Officials: Ian F Tannock, MD, PhD, DSc, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada